CLINICAL TRIAL: NCT01097772
Title: A Clinical Study to Evaluate the Safety and Performance of the TriVascular Ovation™ Abdominal Stent Graft System
Brief Title: TriVascular European Union (EU) Abdominal Stent Graft Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TriVascular, Inc. (Industry)
Responsible Party: Sponsor
Organization: Endologix (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 771-0004
Record Dates: First submitted 2010-03-31; First posted 2010-04-02 (Estimated); Last update posted 2021-06-04 (Actual); Status verified 2021-06

CONDITIONS: Abdominal Aortic Aneurysm
Keywords: abdominal; aortic; aneurysm
MeSH Terms: conditions — Aortic Aneurysm, Abdominal; Aneurysm

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ovation Abdominal Stent Graft System (Other): Implant of Ovation Abdominal Stent Graft System
  Interventions: Device: Implant of Ovation Abdominal Stent Graft System

INTERVENTIONS:
Device: Implant of Ovation Abdominal Stent Graft System — Single occurrence permanent implant of AAA device.

SUMMARY:
A Clinical Study to Evaluate the Safety and Performance of the TriVascular Ovation Abdominal Stent Graft System

DETAILED DESCRIPTION:
A prospective, consecutively enrolling, non-randomized multi center clinical evaluation of the safety and performance of the TriVascular AAA Stent Graft when used in the treatment of patients with Abdominal Aortic Aneurysms (AAA).

ELIGIBILITY:
Inclusion Criteria:

1. Patient is > 18 years of age
2. Patients who are male or non-pregnant female (females of child bearing potential must have a negative pregnancy test prior to enrollment into the study)
3. Patient has signed an Ethics Committee (EC) approved Informed Consent Form
4. Patient is considered by the treating physician to be a candidate for elective open surgical repair of the AAA (i.e., category I, II, or III per American Society of Anesthesiology (ASA) classification; refer to Appendix III: ASA Classification System). ASA category IV patients may be enrolled provided their life expectancy is greater than 1 year.
5. Patient has an infrarenal abdominal aortic aneurysm that meets at least one of the following:

   * Abdominal aortic aneurysm ≥5.0 cm in diameter
   * Aneurysm has increased in size by 0.5 cm in last 6 months.
   * Maximum diameter of aneurysm exceeds 1.5 times the transverse dimension of an adjacent non-aneurysmal aortic segment
6. Patient has patent iliac or femoral arteries that allow endovascular access with the TriVascular AAA device.
7. Patient has a suitable non-aneurysmal proximal aortic neck length of ≥ 7 mm inferior to the most distal renal artery ostium.
8. Patient has a suitable non-aneurysmal distal iliac artery length (seal zone) of ≥10 mm. The resultant repair should preserve patency in at least one hypogastric artery.
9. Patient has a suitable non-aneurysmal proximal aortic neck luminal diameter between 16 and 30 mm.
10. Patient has suitable non-aneurysmal distal iliac luminal diameters between 8 and 20 mm.
11. Patient meets the following anatomic criteria: the distance from the most distal renal artery to most superior internal iliac artery measurement is at least 13 cm.
12. Patient has juxtarenal aortic neck angulation ≤ 60º if proximal neck is ≥10 mm and ≤ 45º if proximal neck is <10 mm.
13. Patient must be willing to comply with all required follow-up exams.

Exclusion Criteria:

1. Patient has a dissecting aneurysm
2. Patient has an acutely ruptured aneurysm
3. Patient has an acute vascular injury
4. Patient has a need for emergent surgery
5. Patient has a known thoracic aortic aneurysm or dissection.
6. Patient has a mycotic aneurysm or has an active systemic infection
7. Patient has unstable angina (defined as angina with a progressive increase in symptoms, new onset at rest or nocturnal angina, or onset of prolonged angina)
8. Patient has had a myocardial infarction (MI) and/or stroke (CVA) within the past 6 months.
9. Patient has a major surgical or interventional procedure planned ≤30 days of the AAA repair.
10. Patient has history of connective tissue disease (e.g., Marfan's or Ehler's-Danlos syndrome).
11. Patient has history of bleeding disorders or refuses blood transfusions.
12. Patient has dialysis dependent renal failure or baseline serum creatinine level >2.0 mg/dl
13. Patient has a known hypersensitivity or contraindication to anticoagulation or contrast media that is not amenable to pre-treatment.
14. Patient has a known allergy or intolerance to polytetrafluoroethylene (PTFE), PEG-based polymers or nitinol.
15. Patient has a body habitus that would inhibit X-ray visualization of the aorta
16. Patient has a limited life expectancy of less than 1 year
17. Patient is currently participating in another investigational device or drug clinical trial
18. Patient has other medical, social or psychological conditions that, in the opinion of the investigator, preclude them from receiving the pre-treatment, required treatment, and post-treatment procedures and evaluations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-03 (Actual); Primary Completion 2010-10-29 (Actual); Study Completion 2015-09-16 (Actual)

PRIMARY OUTCOMES:
The primary safety endpoint is defined as the proportion of subjects who experience a Serious Adverse Event within 30 days of the initial procedure. | 30-Days
  The safety of the TriVascular AAA Stent Graft will be determined by comparing the rate of Serious Adverse Events in the Treatment Group against the rate of Serious Adverse Events in the Control Group within 30 days of the initial procedure.

SECONDARY OUTCOMES:
To evaluate the performance of the TriVascular AAA Stent-Graft System within 30 days of the initial procedure. | 30-Days
  The performance of the TriVascular AAA Stent-Graft System will be determined by comparing the composite success rate in the Treatment Group against an estimated success rate of 80% in the Control Group within 30 days of the initial procedure. The composite success rate is defined as:
  1. Technical Success, defined as successful delivery and deployment of one aortic body and two iliac limbs.
  2. Absence of Type I and III endoleaks
  3. Absence of Rupture
  4. Absence of Conversion to Open Surgical Repair
  5. Freedom from mortality

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Nolte, MD, Principal Investigator — Herz- und Gefässzentrum Bad Bevensen
Locations (7):
- Germany (7):
  - Herz- und Gefässzentrum Bad Bevensen, Bad Bevensen
  - Univeristy Klinik Köln, Cologne
  - Klinikum Dortmund GmbH, Dortmund
  - Cardiovascular Center Frankfurt-Sankt Katherinen, Frankfurt
  - Universitäres Herz und Gefäß Zentrum Hamburg, Hamburg
  - Herzzentrum Leipzig, Leipzig
  - St Franziskus Hospital Munster, Münster

REFERENCES:
- [Derived] Mehta M, Valdes FE, Nolte T, Mishkel GJ, Jordan WD, Gray B, Eskandari MK, Botti C; A Pivotal Clinical Study to Evaluate the Safety and Effectiveness of the Ovation Abdominal Stent Graft System Investigators. One-year outcomes from an international study of the Ovation Abdominal Stent Graft System for endovascular aneurysm repair. J Vasc Surg. 2014 Jan;59(1):65-73.e1-3. doi: 10.1016/j.jvs.2013.06.065. Epub 2013 Aug 24. PMID 23978572